CLINICAL TRIAL: NCT05107154
Title: iCARE 2.0: A Pilot Intervention of Dialectical Behavioural Therapy for Youth With Type 2 Diabetes.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Brandy Wicklow (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor-Investigator, Dr. Brandy Wicklow, Principle Investigator, University of Manitoba
Organization: University of Manitoba (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: B2021:079
Record Dates: First submitted 2021-10-19; First posted 2021-11-04 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Diabetes Mellitus Type 2, Childhood-Onset
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dialectical Behavioural Therapy (Experimental): Participants randomized to the Dialectical Behavioural Therapy (DBT) skills training intervention will receive a 90-minute DBT skills training session every week for 16 weeks total. The sessions will be facilitated by a health practitioner supervised by a clinical health psychologist with expertise in program development and DBT-adaptations for a variety of populations. Sessions for Pilot 1 will be delivered via Zoom HealthCare and in person if allowable. In-person sessions would be delivered at the Children's Hospital Research Institute of Manitoba. Pilot 2 will be adapted to address any additional needs uncovered through he qualitative assessment of Pilot 1. Traditional medicine components will be developed within the first 2 years of the grant by Indigenous researchers, patient and parent advisors, elders, and community advisory groups. These elements will be offered as an encouraged, yet optional component (additional modules) within the 16-week DBT intervention in Pilot 2.
  Interventions: Behavioral: Dialectical Behavioural Therapy
- Control (No Intervention): Participants randomized to the control arm will receive standard medical care and clinical follow-up. Controls will be offered DBT after completion of Pilot 1 and 2. Participation will be optional.

INTERVENTIONS:
Behavioral: Dialectical Behavioural Therapy — DBT skills training is organized into 5 specific modules designed to support skills needed to control emotional reactivity, including: Mindfulness, Distress Tolerance, Walking the Middle Path (a family-based module developed by our co-investigators specifically for teens), Emotion Regulation, and Interpersonal Effectiveness.
  Arms: Dialectical Behavioural Therapy

SUMMARY:
In partnership with youth, parents, and community members the investigators have co-developed a program of research designed to address the substantial health disparities faced by First Nations children and families, and the calls to action from the Truth and Reconciliation Report. Specifically; the investigators aim to address the high rates of kidney disease in Indigenous children living with Type 2 Diabetes (T2D), by identifying and understanding the root causes for progression of kidney disease and working together to build an evidenced based, novel therapy for diabetes that focuses on mindfulness, personal strengths and incorporates traditional medicine practices that are meaningful to patients.

The investigators have planned 2 pilots in order to address the uncertainties surrounding the planning of a larger definitive trial and allow adequate engagement and building of a meaningful traditional medicine component. These pilots will inform the development of a co-designed, feasible, and embraced Dialectical Behavioural Therapy (DBT) skills training and traditional teachings intervention, which is adequately powered to examine effectiveness on outcomes such as mental wellness, medication adherence, and improved glycemic control and renal function.

Research Aims: 1. Determine the recruitment, enrollment and adherence rates to the intervention. 2. Evaluate acceptability of the intervention using traditional qualitative methods and Indigenous world view methodology 3. Determine the estimated effect size required to power a large-scale DBT randomized control trial for the outcomes quality of life (primary), glycemic control and albuminuria (secondary).

Study Hypotheses: 1. The investigators hypothesize that a DBT intervention will be feasible on a local and National Platform and will be acceptable and embraced by youth with T2D as an important component of their management plan. 2. The investigators hypothesize that the additional of traditional medicine elements will increase the acceptability and adherence to DBT for Indigenous children.

DETAILED DESCRIPTION:
The investigators will conduct a quasi-experimental trial with a small sample of adolescents and one family member to participate in group-based Dialectical Behavioural Therapy (DBT) or be randomized to a control arm. Pre-measures, post-measures, and 3-month follow up measures will be collected on DBT participants and control participants. Participants receiving DBT and parents/guardian of the DBT participants will also be asked to complete 1-on-1 qualitative interviews after the 16-week program is finished. Pilot 1 will consist of group-based DBT and Pilot 2 will consist of group-based DBT with an optional component which incorporates traditional Indigenous medicines and knowledge. Pilot 2 will be built with Indigenous scholars and elders and will be submitted as an amendment to the University of Manitoba Research Ethics Board when appropriate consultation has been completed. We are only requesting approval for Pilot 1 at this time.

Screening, Enrolment and Intervention Assignment: Research assistants will recruit participants from the Diabetes Education Resource for Children and Adolescents, located in the Community Services Building at the Health Science Center in Winnipeg, Manitoba. Participants currently enrolled in the iCARE Cohort, who have consented to be contacted about future studies and who meet eligibility requirements will also be approached to share information about this study. Interested participants will be screened utilizing a number of questionnaires and self-report measures in person (if allowable), via telephone, or on REDCap

Pilot 1 will be completed virtually through Zoom HealthCare.

The main outcome measures for the pilot trials were selected to inform the feasibility and sample size required for a larger RCT on a national scale. These include recruitment rates, retention rates, adherence to the intervention, retention for follow-up measurements, and satisfaction with the intervention. The investigators will also assess youth and parent experiences and perceptions of the intervention using inductive qualitative research upon completion of the 16-week trial.

The proposed intervention is mental health support intervention, therefore it does not include medication therapy or devices. The program is being delivered by trained clinical psychologist/psychology students.

Debriefing occurs throughout the intervention to assess for significant mental distress (including but not limited to weekly check-ins). Individual mental health concerns will be dealt with with as they arise. If at any point during the clinical research, clinicians judge the program is no longer beneficial or actively detrimental to an individual's health and wellbeing, the team has the right to end services and provide referrals and support for other treatment models.

Adverse events (AE) will be collected to document unfavorable changes in current health status of the research participant or any incident, experience or outcome that suggests that the research may place participants or others at a greater risk of harm (including physical, psychological, economic or social harm). The AE's that will be reported will include complications from the blood draw (syncopal episode, infection, excessive bleeding requiring medical attention), or events that could be related to completing the mental health questionnaires (emergency visit or crisis resource utilization or hospitalization for suicidal ideation, attempt). All deaths, regardless of cause will also be recorded for participants active in the study.

Sample Size Assessment

Sample size analysis showed that a full-scale trial would require 150 subjects (using a standardized effect size of 0.4 scale change in the self reported quality of life for an individual). The investigators chose to use 10% of this for each pilot (n=15) and added a control arm of n=15 for each pilot as well.

Quantitative Analytic Plan

For feasibility outcomes the investigators will be looking for a minimum 70% adherence (i.e. completing 11/16 sessions) in order to properly test the study hypothesis with a larger trial. A minimum 85% retention rate at follow-up (i.e. percentage of randomized participants that provide outcome measures at follow-up) is needed to protect the original randomization. For estimated effect size of the intervention the investigators will test for group-wise differences in the outcome measures using a repeated measures mixed effects regression model with a random subject effect to account for the within-subject correlations and repeated measures design with outcomes assessed at baseline and 16 weeks. Fixed effects will include treatment, time, and their interaction. An intention to treat strategy will be adopted for the final analysis. The analysis will be underpowered to test for effects for boys and girls separately, however sex as an interaction term in the analysis will be added.

Qualitative Analytic Plan

Youth & parents/guardian from the DBT intervention arm of both pilot studies (n = 30) will participate in end-point semi-structured interviews of 45-minute duration, guided by Interpretive Description methodology. Interpretive description is a non-categorical applied research approach that seeks to generate understanding of clinically relevant phenomena in relation to its local context. An investigator (M.A) with extensive qualitative research experience will conduct all interviews. Interviews will be conducted via Zoom HealthCare or in-person if allowable. Questions will focus on perceptions of intervention delivery (e.g., duration, dose, timing, interventionist); content (e.g., domains); experiences - including emotional and cognitive responses; and intervention acceptability.

Audio recorded data will be transcribed verbatim and managed using NVivo software (version 1.0). Data from the first three transcripts will inform development of a coding framework which will be applied to subsequent interviews and iteratively revised upon identification of new conceptually distinct codes. Codes will be grouped into thematic clusters with supporting narrative excerpts. Thematic data will be used to refine what the investigators determine as modifiable domains of DBT.

ELIGIBILITY:
Inclusion Criteria:

* Thirty (30) youths (ages 14-22 years old) living with youth onset T2D will be recruited to participate in Pilot 1, fifteen (15) youths, and one caregiver, will be randomized to receive DBT and fifteen (15) adolescents will be randomized to a control group.
* An additional thirty youths (14-22 years old) will be recruited to participate in Pilot 2.

Exclusion Criteria:

* Diabetes not diagnosed as type 2 diabetes including: type 1 diabetes, genetic diabetes, cystic fibrosis diabetes, diabetes secondary to medication use.
* Ever cancer
* Other chronic illness associated with systemic inflammation (ex. Juvenile rheumatoid arthritis, Crohn's disease)
* Active psychotic disorder
* Past year suicide attempt or an active plan
* Self-reported substance/alcohol use disorder in past (1 year)
* Patient and/or caregiver unable or unwilling to provide voluntary informed assent/consent
* Currently pregnant (eligible at 3 months post-partum)
* Exclusion criteria would include significant self-harm behaviour and substance abuse, which would impair affective participation in a DBT group setting based on clinical judgement.

Ages: 14 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-11-21 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Study Feasibility | 1 year per pilot
  Determine the recruitment, enrollment, and adherence rates to the intervention.
Study Acceptability | 1 year per pilot
  Participant semi-structured interviews will be conducted to generate understanding of the patient experience, including elements of the intervention that were most useful, and elements requiring modification informing needed adaptations for future studies.
Pediatric Quality of Life (PedsQL) | 1 year per pilot
  The Pediatric Quality of Life (PedsQL - Teen/Young Adult) questionnaire will be used to determine the impact Dialectical Behavioural Therapy (DBT) has on pediatric quality of life. Results will also be used to determine the estimated effect size required to power a large-scale DBT randomized control trial.

SECONDARY OUTCOMES:
Albuminuria | 1 year per pilot
  Albumin:creatinine ratio (ACR) testing will be used to determine the impact Dialectical Behavioural Therapy (DBT) has on albuminuria (>2.0mg/mmol, 1st morning urine collection). results will also be used to determine the estimated effect size required to power a large-scale DBT randomized control trial
Glycemic Control | 1 year pilot
  Glycemic control will be measured by Hemoglobin A1c and changes pre-post will be measured to identify any impact of the intervention on diabetes control.

CONTACTS AND LOCATIONS:
Overall Officials: Brandy Wicklow, MD MSc, Principal Investigator — University of Manitoba
Locations (2):
- Canada (2):
  - Clinic Y, Health Sciences Centre, Winnipeg, Manitoba
  - Diabetes Education Resource Centre for Adolescents Clinic, Health Sciences Centre, Winnipeg, Manitoba

IPD SHARING:
Plan to Share IPD: No